CLINICAL TRIAL: NCT00484328
Title: Ribavirin, Its Dosing Regime
Acronym: Ribados
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Prof. A.Bast, Maastricht University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MEC-07-3-007
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2011-07

CONDITIONS: Hepatitis C
Keywords: hepatitis C; Ribavirin; Dosage; Pharmacokinetics
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ribavirin
- 2 (Experimental)
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — different dosing regimes of Ribavirin

SUMMARY:
The purpose of this study is to determine if the medicines for chronic hepatitis C can be taken once daily, instead of twice daily.

DETAILED DESCRIPTION:
The standard treatment of patients with chronic hepatitis C infection (HCV) is treatment with ribavirin. Actually, the compliance (2x daily) seems to be a problem. To increase patients' compliance, it is investigated if the total dose of ribavirin can be taken once daily.

The pharmacokinetics of ribavirin at different dosage regimes is investigated.

ELIGIBILITY:
Inclusion Criteria:

* anti-HCV positivity > 6 months
* Positive HCV-RNA genotype 1 or 4
* Liver biopsy within one year before the start of therapy
* Intention to be treated and participate treatment
* body weight at or above 75 kg

Exclusion Criteria:

* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetics of ribavirin at different dosage regimes, measured by the area under the curve of the concentration-time graph | within 24 weeks after enrollment

SECONDARY OUTCOMES:
The tolerability of the treatment at different dosage regimes of ribavirin | 24 weeks of treatment
The antioxidant capacity in plasma and erythrocytes at different dosing regimes | 24 weeks of treatment
The effect of ribavirin on the hemolysis | 24 weeks of treatment
The pharmacokinetics of ribavirin in erythrocytes in the different dosing regimes | 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aalt Bast, Prof.Dr., Principal Investigator — Maastricht University
Locations (1):
- University of Maastricht, Maastricht, Netherlands